CLINICAL TRIAL: NCT03865446
Title: A PHASE 1, OPEN-LABEL, SINGLE-DOSE, PARALLEL-GROUP STUDY TO EVALUATE THE PLASMA PHARMACOKINETICS AND SAFETY OF DACOMITINIB IN PARTICIPANTS WITH SEVERELY IMPAIRED HEPATIC FUNCTION RELATIVE TO PARTICIPANTS WITH NORMAL HEPATIC FUNCTION
Brief Title: Evaluate Severe Hepatic Impairment on Dacomitinib PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A7471058
Record Dates: First submitted 2019-02-07; First posted 2019-03-06 (Actual); Results first posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-10

CONDITIONS: Severe Hepatic Impairment
Keywords: Pharmacokinetics; Dacomitinib; Hepatic Impairment
MeSH Terms: interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Dacomitinib) (Experimental): severe hepatic impairment group
  Interventions: Drug: Dacomitinib
- Cohort 2 (Dacomitinib) (Experimental): normal hepatic function
  Interventions: Drug: Dacomitinib

INTERVENTIONS:
Drug: Dacomitinib — anti-cancer agent
  Other Names: PF-00299804; VIZIMPRO

SUMMARY:
This is a post approval requirement to study the effect of severe hepatic impairment on the pharmacokinetics of dacomitinib.

DETAILED DESCRIPTION:
This is a Phase 1, open label, parallel group study to investigate the effect of severe hepatic impairment on the plasma PK, safety and tolerability after a single oral 30 mg dose of dacomitinib under fasted conditions.

Approximately 18 participants will be enrolled into the study to ensure at least 6 PK evaluable (having data for estimating primary PK parameters for dacomitinib) participants in each cohort.

ELIGIBILITY:
Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Male and/or female participants of non childbearing potential must be 18 to 75 years of age, inclusive, at the time of signing the informed consent document (ICD).
2. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

   Weight:
3. Body mass index (BMI) of 17.5 to 40 kg/m2; and a total body weight >50 kg (110 lb).
4. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Any condition possibly affecting drug absorption (eg, gastrectomy).
2. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or IP administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
3. History of or current positive results for human immunodeficiency virus (HIV).
4. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of IP used in this study (whichever is longer).
5. Hypersensitivity to dacomitinib or its excipients.
6. A positive urine drug test. Participants with severe hepatic impairment (Cohort 1) will be eligible to participate if their urine drug test is positive with a drug for a prescribed condition that is not expected to interfere with the PK of dacomitinib.
7. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
8. History of sensitivity to heparin or heparin induced thrombocytopenia.
9. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
10. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Sponsor employees, including their family members, directly involved in the conduct of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2019-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Investigational Drug Services (IDS) University of Miami Hospitals and Clinics, Research Pharmacy, Miami, Florida
  - University of Miami Division of Clinical Pharmacology, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Piscitelli J, Chen J, LaBadie RR, Salageanu J, Chung CH, Tan W. The Effect of Hepatic Impairment on the Pharmacokinetics of Dacomitinib. Clin Drug Investig. 2022 Mar;42(3):221-235. doi: 10.1007/s40261-022-01125-x. Epub 2022 Feb 23. PMID 35195881
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A7471058

RESULTS

PARTICIPANT FLOW:
Groups:
- Severe Hepatic Impairment: Participants with severe hepatic impairment received a single oral dose of dacomitinib 30 milligram (mg) tablet on Day 1 and were followed up to a maximum of 35 days for safety.
- Normal Hepatic Function: Participants with normal hepatic function received a single oral dose of dacomitinib 30 mg tablet on Day 1 and were followed up to a maximum of 35 days for safety.
Period: Overall Study
Arm/Group | Severe Hepatic Impairment | Normal Hepatic Function
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants assigned to dacomitinib and who take 1 dose of dacomitinib.
Groups:
- Severe Hepatic Impairment: Participants with severe hepatic impairment received a single oral dose of dacomitinib 30 mg tablet on Day 1 and were followed up to a maximum of 35 days for safety.
- Total: Total of all reporting groups
Arm/Group | Severe Hepatic Impairment | Normal Hepatic Function | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (6.82) | 59.0 (5.37) | 59.5 (5.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Dacomitinib
Description: Cmax of Dacomitinib was analyzed.
Time Frame: Pre-dose and 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216 and 264 hours post dose on Day 1
Population: Pharmacokinetic (PK) population included all participants who took one dose of dacomitinib and had at least one dacomitinib plasma PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Severe Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 8 | 8
nanogram per milliliter | 9.673 (35) | 7.389 (63)
Statistical Analysis 1: Comparison: Severe Hepatic Impairment vs Normal Hepatic Function; Test type: Other; Geometric Means Ratio = 130.91, 90% CI 2-sided [86.03 to 199.22] — The model was an analysis of variance (ANOVA) model with unequal variance assumption and hepatic impairment group as fixed effect. Values were back-transformed from the log scale

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinite Time (AUCinf) of Dacomitinib
Description: AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf).
Time Frame: Pre-dose and 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216 and 264 hours post dose on Day 1
Population: PK population included all participants who took one dose of dacomitinib and had at least one dacomitinib plasma PK parameters of primary interest. Here, 'Overall Number of Participants Analyzed' = participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Severe Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 8 | 7
nanogram*hour per milliliter | 735.0 (37) | 703.9 (48)
Statistical Analysis 1: Comparison: Severe Hepatic Impairment vs Normal Hepatic Function; Test type: Other; Geometric Means Ratio = 104.41, 90% CI 2-sided [72.12 to 151.16] — The model was an ANOVA model with unequal variance assumption and hepatic impairment group as fixed effect. Values are back-transformed from the log scale

3. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Laboratory abnormalities included hematology- Erythrocyte mean corpuscular hemoglobin: less than (<) 0.9 *lower limit of normal (LLN), platelets: < 0.5* LLN, leukocytes: < 0.6* LLN, lymphocytes: < 0.8* LLN, eosinophils: greater than (>) 1.2* lower limit of normal (ULN), partial thromboplastin time (PTT): > 1.1* ULN, prothrombin time: > 1.1* ULN, Prothrombin Intl. normalized ratio: > 1.1* ULN, clinical chemistry- bilirubin: > 1.5* ULN, protein: < 0.8* LLN, albumin: < 0.8* LLN, urinalysis- urine protein: greater than or equal to (>=) 1, urine hemoglobin: >= 1, urobilinogen: >= 1, urine erythrocytes: >= 20.
Time Frame: Baseline up to Day 7
Population: Safety population included all participants assigned to dacomitinib and who took one dose of dacomitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 8 | 8
Participants | 8 | 5

4. Secondary Outcome: Number of Participants With Physical Examination Abnormalities
Description: Height and weight were measured to calculate body mass index abnormality.
Time Frame: Baseline up to Day 7
Population: Safety population included all participants assigned to dacomitinib and who took one dose of dacomitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With Vital Sign Parameters Meeting Criteria of Potential Clinical Concern
Description: Systolic blood pressure, diastolic blood pressure and pulse rate were evaluated for examination of vital signs. Criteria for potential concern in absolute values of vital sign: pulse rate: <40 beats per minute (bpm), >120 beats per minute; supine diastolic blood pressure: <50 millimeter of mercury (mm Hg); supine systolic blood pressure: <90 mm Hg. Criteria for potential concern in change from baseline in vital sign values: supine diastolic blood pressure: greater than or equal to >= 30 mm Hg increase or decrease from baseline; supine diastolic blood pressure: >=20 mm Hg increase or decrease from baseline. Only participants with vital sign parameters meeting criteria of potential clinical concern are reported.
Time Frame: Baseline up to Day 7
Population: Safety population included all participants assigned to dacomitinib and who took one dose of dacomitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 8 | 8
Participants
  Increase in systolic blood pressure | 1 | 0
  Increase in diastolic blood pressure | 0 | 1

6. Secondary Outcome: Number of Participants With ECG Parameters Meeting Criteria of Potential Clinical Concern
Description: ECG parameters RR interval, PR interval, QRS interval, QT interval, QTC interval, QTCB, QTCF and heart rate were measured. Criteria of potential concern for absolute values: PR interval: >=300 milliseconds; QRS interval >=140 milliseconds; QT interval: >=500 milliseconds; QTCF (Fridericia's correction formula) : >= 450 to < 480 milliseconds, >=480 to <500 milliseconds, >=500 milliseconds. Criteria of potential concern for change from baseline values: PR interval: when baseline is >200 millisecond- change >=25%, when baseline <200 milliseconds- change >=50%; QRS interval: change >= 50%; QTCF: change >=30 to <60, change >=60. In this outcome measure, participants meeting the criteria of potential concern for any of the ECG parameters are reported.
Time Frame: Baseline up to Day 7
Population: Safety population included all participants assigned to dacomitinib and who took one dose of dacomitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 8 | 8
Participants | 1 | 0

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events. A treatment emergent AE was defined as an event that emerged during the treatment period (Up to Day 35) that was absent before treatment, or worsened during the treatment period relative to the pretreatment state.
Time Frame: Baseline up to Day 35
Population: Safety population included all participants assigned to dacomitinib and who took one dose of dacomitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 8 | 8
Participants
  AEs | 0 | 0
  SAEs | 0 | 0

8. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Treatment-emergent are events between first dose of study drug and up to 35 days after first dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Dacomitinib was assessed by the investigator.
Time Frame: Baseline up to Day 35
Population: Safety population included all participants assigned to dacomitinib and who took one dose of dacomitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Hepatic Impairment | Normal Hepatic Function
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 35
Arm/Group | Severe Hepatic Impairment | Normal Hepatic Function
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/46/NCT03865446/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT03865446/SAP_001.pdf